CLINICAL TRIAL: NCT06261671
Title: Antioxidants-enriched Single-step vs Global Total Single-step Embryo Culture Media: Effect on Blastocyst Euploidy Rates.
Brief Title: Effect of Antioxydant-enriched Media on Blastocyst Euploidy Rates.
Acronym: GX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2312-ABU-028-VF
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Infertility; In Vitro Fertilization
Keywords: Intracytoplasmic sperm injection; Pre - implanttaion genetic diagnosis for aneuploidy; Antioxydante; Culture media; Embryo development; Euploidy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: A randomization list (indicating Gx Media Vitrolife or GT Coopersurgical) will be used to verify to which group the first half of oocytes will be allocated to. In case an odd number of oocytes is present, one extra oocyte is allocated to the group as indicated by the randomization list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: antioxidants-enriched culture medium (Gx) (Active Comparator): Blastocyst exposed to antioxidants-enriched culture medium (Gx) in continuous culture conditions, without refreshment on day 3. A refreshment of the media will be done on D5 in both groups.
  Interventions: Drug: antioxidants-enriched culture medium (Gx)
- Group 2: Global total one step media (GT) (Active Comparator): Blastocyst exposed to Global total one step media (GT) in continuous culture conditions, without refreshment on day 3. A refreshment of the media will be done on D5 in both groups.
  Interventions: Drug: antioxidants-enriched culture medium (Gx)

INTERVENTIONS:
Drug: antioxidants-enriched culture medium (Gx) — Blastocyst will be in continuous culture conditions (parallel antioxidants-enriched culture medium (Gx) and Global total one step media (GT) without refreshment on day 3. A refreshment of the media will be done on D5 in both groups.
  Other Names: Global total one step media (GT)

SUMMARY:
One of the most sensible factors in IVF culture conditions is the susceptibility of gametes and embryos to an induced increase in reactive oxidative species (ROS) caused by the artificial environment. This study aims to evaluate the impact of using antioxidant-supplemented media during culture to evaluate embryo ploidy rates in a prospective randomized trial using sibling oocytes.

DETAILED DESCRIPTION:
Improvements in culture conditions is an ongoing process in IVF due to, on one hand, the still lack of knowledge on human embryonic development, and, on the other hand, the frequent need for repeated IVF cycles to achieve an 'implantable' embryo. The main factor for optimizing conditions of an embryo to develop is its microenvironment, mainly the culture media used. One of the most sensible factors in IVF culture conditions is the susceptibility of gametes and embryos to an induced increase in reactive oxidative species (ROS) caused by the artificial environment, as it has been extensively shown in animal models and to a certain extent in humans.

A primordial step for improvement is to alleviate an increase in ROS during embryo development. This can be manipulated by means of utilizing a culture media with supplements that can serve as scavengers, leading to an equilibrium between oxidation and reduction of ROS during the culture period. So far, the produced culture media contain low concentrations of limited additives involved in anti-oxidative stress. Recently, a culture medium containing an implementation in higher doses of distinctive elements known to clearly serve as cellular scavengers has been formulated. However, very few human IVF studies have been performed up to date. Our research intends to investigate the incorporation of antioxidant-rich culture media into IVF practices with the primary objective of analyzing its impact on embryo euploidy, as well as the previous culture steps including fertilization and blastocyst developmental rates. This study aims to evaluate the impact of using antioxidant-supplemented media during culture to evaluate embryo ploidy rates in a prospective randomized trial using sibling oocytes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing assisted reproductive technology cycles when ICSI is indicated.
* Patients when Iin vitto fertilization (IVF) is also performed will be included as far as there are enough oocytes for ICSI randomization. However, IVF oocytes will not be used for the study.
* Maternal age 18-43 years old.
* PGT-A cycles with only trophectoderm biopsies on day 5/6/7.
* Patients with more than 6 COCs expected for ICSI.
* Body mass index <35.
* Fresh and frozen ejaculated sperm.

Exclusion Criteria:

* PGT-M cycles
* Fresh and frozen testicular sperm.

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blastocyst ploidy is determined after a biopsy of trophectoderm cells, taken from the blastocyst on day 5, 6 or 7 from development. The following outcomes are possible: • Normal • Abnormal • No result/Inconclusive • Low or high Mosaic | 1 year
  Ploidy rate is calculated by dividing the number of normal embryos by the number of blastocysts biopsied in the group.

SECONDARY OUTCOMES:
Cycle ploidy rate: the number of euploid embryos in the group Blastocyst quality at the time of biopsy based on modified Gardner's criteria. Usable blastocyst rate per group and per day of biopsy (day 5, 6, 7) | 1 year
  Ploidy rate is calculated by dividing the number of normal embryos by the number of blastocysts biopsied in the group.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, Study Director — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meldrum DR, Casper RF, Diez-Juan A, Simon C, Domar AD, Frydman R. Aging and the environment affect gamete and embryo potential: can we intervene? Fertil Steril. 2016 Mar;105(3):548-559. doi: 10.1016/j.fertnstert.2016.01.013. Epub 2016 Jan 23. PMID 26812244
- [Background] von Mengden L, Klamt F, Smitz J. Redox Biology of Human Cumulus Cells: Basic Concepts, Impact on Oocyte Quality, and Potential Clinical Use. Antioxid Redox Signal. 2020 Mar 10;32(8):522-535. doi: 10.1089/ars.2019.7984. PMID 31861967
- [Background] Ruder EH, Hartman TJ, Blumberg J, Goldman MB. Oxidative stress and antioxidants: exposure and impact on female fertility. Hum Reprod Update. 2008 Jul-Aug;14(4):345-57. doi: 10.1093/humupd/dmn011. Epub 2008 Jun 4. PMID 18535004
- [Background] Chambers GM, Dyer S, Zegers-Hochschild F, de Mouzon J, Ishihara O, Banker M, Mansour R, Kupka MS, Adamson GD. International Committee for Monitoring Assisted Reproductive Technologies world report: assisted reproductive technology, 2014dagger. Hum Reprod. 2021 Oct 18;36(11):2921-2934. doi: 10.1093/humrep/deab198. PMID 34601605
- [Background] Halliwell B, Aruoma OI. DNA damage by oxygen-derived species. Its mechanism and measurement in mammalian systems. FEBS Lett. 1991 Apr 9;281(1-2):9-19. doi: 10.1016/0014-5793(91)80347-6. PMID 1849843
- [Background] Kehrer JP, Lund LG. Cellular reducing equivalents and oxidative stress. Free Radic Biol Med. 1994 Jul;17(1):65-75. doi: 10.1016/0891-5849(94)90008-6. PMID 7959167
- [Background] Aitken RJ. Impact of oxidative stress on male and female germ cells: implications for fertility. Reproduction. 2020 Apr;159(4):R189-R201. doi: 10.1530/REP-19-0452. PMID 31846434
- [Background] Ruder EH, Hartman TJ, Goldman MB. Impact of oxidative stress on female fertility. Curr Opin Obstet Gynecol. 2009 Jun;21(3):219-22. doi: 10.1097/gco.0b013e32832924ba. PMID 19469044
- [Background] Agarwal A, Said TM. Role of sperm chromatin abnormalities and DNA damage in male infertility. Hum Reprod Update. 2003 Jul-Aug;9(4):331-45. doi: 10.1093/humupd/dmg027. PMID 12926527
- [Background] Lian HY, Gao Y, Jiao GZ, Sun MJ, Wu XF, Wang TY, Li H, Tan JH. Antioxidant supplementation overcomes the deleterious effects of maternal restraint stress-induced oxidative stress on mouse oocytes. Reproduction. 2013 Oct 21;146(6):559-68. doi: 10.1530/REP-13-0268. Print 2013 Dec. PMID 24043846
- [Background] Kiani-Esfahani A, Bahrami S, Tavalaee M, Deemeh MR, Mahjour AA, Nasr-Esfahani MH. Cytosolic and mitochondrial ROS: which one is associated with poor chromatin remodeling? Syst Biol Reprod Med. 2013 Dec;59(6):352-9. doi: 10.3109/19396368.2013.829536. Epub 2013 Aug 22. PMID 23968144
- [Background] Lu J, Wang Z, Cao J, Chen Y, Dong Y. A novel and compact review on the role of oxidative stress in female reproduction. Reprod Biol Endocrinol. 2018 Aug 20;16(1):80. doi: 10.1186/s12958-018-0391-5. PMID 30126412
- [Background] Agarwal A, Rana M, Qiu E, AlBunni H, Bui AD, Henkel R. Role of oxidative stress, infection and inflammation in male infertility. Andrologia. 2018 Dec;50(11):e13126. doi: 10.1111/and.13126. PMID 30569652
- [Background] Guerin P, El Mouatassim S, Menezo Y. Oxidative stress and protection against reactive oxygen species in the pre-implantation embryo and its surroundings. Hum Reprod Update. 2001 Mar-Apr;7(2):175-89. doi: 10.1093/humupd/7.2.175. PMID 11284661
- [Background] Hardy MLM, Day ML, Morris MB. Redox Regulation and Oxidative Stress in Mammalian Oocytes and Embryos Developed In Vivo and In Vitro. Int J Environ Res Public Health. 2021 Oct 29;18(21):11374. doi: 10.3390/ijerph182111374. PMID 34769890
- [Background] Carbone MC, Tatone C, Delle Monache S, Marci R, Caserta D, Colonna R, Amicarelli F. Antioxidant enzymatic defences in human follicular fluid: characterization and age-dependent changes. Mol Hum Reprod. 2003 Nov;9(11):639-43. doi: 10.1093/molehr/gag090. PMID 14561807
- [Background] Mauchart P, Vass RA, Nagy B, Sulyok E, Bodis J, Kovacs K. Oxidative Stress in Assisted Reproductive Techniques, with a Focus on an Underestimated Risk Factor. Curr Issues Mol Biol. 2023 Feb 3;45(2):1272-1286. doi: 10.3390/cimb45020083. PMID 36826028
- [Background] Pigeolet E, Corbisier P, Houbion A, Lambert D, Michiels C, Raes M, Zachary MD, Remacle J. Glutathione peroxidase, superoxide dismutase, and catalase inactivation by peroxides and oxygen derived free radicals. Mech Ageing Dev. 1990 Feb 15;51(3):283-97. doi: 10.1016/0047-6374(90)90078-t. PMID 2308398
- [Background] Van Montfoort APA, Arts EGJM, Wijnandts L, Sluijmer A, Pelinck MJ, Land JA, Van Echten-Arends J. Reduced oxygen concentration during human IVF culture improves embryo utilization and cumulative pregnancy rates per cycle. Hum Reprod Open. 2020 Jan 22;2020(1):hoz036. doi: 10.1093/hropen/hoz036. eCollection 2020. PMID 31989044
- [Background] Truong T, Gardner DK. Antioxidants improve IVF outcome and subsequent embryo development in the mouse. Hum Reprod. 2017 Dec 1;32(12):2404-2413. doi: 10.1093/humrep/dex330. PMID 29136144
- [Background] Bedaiwy M, Agarwal A, Said TM, Goldberg JM, Sharma RK, Worley S, Falcone T. Role of total antioxidant capacity in the differential growth of human embryos in vitro. Fertil Steril. 2006 Aug;86(2):304-9. doi: 10.1016/j.fertnstert.2006.01.025. Epub 2006 Jun 12. PMID 16769062
- [Background] Gardner DK, Kuramoto T, Tanaka M, Mitzumoto S, Montag M, Yoshida A. Prospective randomized multicentre comparison on sibling oocytes comparing G-Series media system with antioxidants versus standard G-Series media system. Reprod Biomed Online. 2020 May;40(5):637-644. doi: 10.1016/j.rbmo.2020.01.026. Epub 2020 Feb 5. PMID 32299733
- [Background] Lan KC, Lin YC, Chang YC, Lin HJ, Tsai YR, Kang HY. Limited relationships between reactive oxygen species levels in culture media and zygote and embryo development. J Assist Reprod Genet. 2019 Feb;36(2):325-334. doi: 10.1007/s10815-018-1363-6. Epub 2018 Nov 10. PMID 30415468